## **INFORMED CONSENT FORM**

Project title:

Determination of DNA repair products in urine after UV irradiation of the skin

November 13, 2020

| INIEGRMED | CONSENT FOR | DARTICIDATION IN | I RESEARCH PROJECT |
|-----------|-------------|------------------|--------------------|

Titel:

## Determination of DNA repair products in urine after UV irradiation of the skin

## Statement from the subject:

I have received written and oral information and I know enough about the purpose, method, advantages and disadvantages of saying yes to participating. I know that participating is voluntary and that I can always withdraw my consent without losing my current or future rights to treatment. I consent to participate in the research project. I have received a copy of this consent sheet as well as a copy of the written information about the project for my own use.

If, during the course of the experiment, significant information about my state of health emerges, I would like information about this:

Yes: \_\_\_\_\_\_

No: \_\_\_\_\_

After finishing the experiment, I wish \_\_\_\_\_(tick this) / I wish not\_\_\_\_\_(tick this) to be informed about the achived results. This information is sent to my population registered address.

Name: \_\_\_\_\_\_

Date: \_\_\_\_\_\_ Signature: \_\_\_\_\_\_

Statement from principle investigator:

I declare that oral information about the project has been provided, written information has been provided and there is consent for the subject to participate.

Name: \_\_\_\_\_\_\_

Date: \_\_\_\_\_\_ Signature: \_\_\_\_\_\_